CLINICAL TRIAL: NCT00953056
Title: A Double-Blind, Randomized, Placebo-Controlled, Safety and Tolerability Study of Live Pentavalent Human-Bovine Reassortant Rotavirus Vaccine in Chinese Healthy Adults, Children and Infants
Brief Title: A Study of V260 in Healthy Chinese Adults, Children and Infants (V260-028)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V260-028; 2009_627
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2011-04-15 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Rotavirus Gastroenteritis
MeSH Terms: interventions — Rotavirus Vaccines; RotaTeq

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort I - RotaTeq™, Adults (Experimental): Adults randomized to receive a single dose of RotaTeq™.
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent
- Cohort I - Placebo, Adults (Placebo Comparator): Adults randomized to receive a single dose of matching placebo to RotaTeq™.
  Interventions: Biological: Comparator: Placebo
- Cohort II - RotaTeq™, Children (Experimental): Children randomized to receive a single dose of RotaTeq™.
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent
- Cohort II - Placebo, Children (Placebo Comparator): Children randomized to receive a single dose of matching placebo to RotaTeq™.
  Interventions: Biological: Comparator: Placebo
- Cohort III - RotaTeq™, Infants (Experimental): Infants randomized to receive 3 doses of RotaTeq™.
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent
- Cohort III - Placebo, Infants (Placebo Comparator): Infants randomized to receive 3 doses of matching placebo to RotaTeq™.
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — Single 2.0 mL dose V260 (RotaTeq™) administered orally at enrollment.
  The 2-mL vaccine consists of an oral solution of 5 live human-bovine reassortant rotaviruses.
  Other Names: V260, RotaTeq™
  Arms: Cohort I - RotaTeq™, Adults; Cohort II - RotaTeq™, Children
Biological: Comparator: Placebo — Single 2.0 mL dose of matching placebo to RotaTeq™ administered orally at enrollment.
  Arms: Cohort I - Placebo, Adults; Cohort II - Placebo, Children
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent — Three 2.0 mL doses of RotaTeq™ administered orally at 3 separate visits scheduled 28 to 70 days apart. The third dose was administered by 32 weeks of age.
  The 2-mL vaccine consists of an oral solution of 5 live human-bovine reassortant rotaviruses.
  Other Names: V260, RotaTeq™.
  Arms: Cohort III - RotaTeq™, Infants
Biological: Comparator: Placebo — Three 2.0 mL doses of matching placebo to RotaTeq™ administered orally at 3 separate visits scheduled 28 to 70 days apart. The third dose was administered by 32 weeks of age.
  Arms: Cohort III - Placebo, Infants

SUMMARY:
This study will assess the safety and tolerability of RotaTeq™ (V260) in the healthy Chinese populations. Approximately 144 participants will be enrolled and equally stratified into three age cohorts, Cohort I ages 19-47 years, Cohort II ages 2-6 years, and Cohort III ages 6-12 weeks. Randomization ratio is 1:1 in each cohort. The study will be conducted sequentially, participants in Cohort I then Cohort II receiving 1 dose of, and then participants in Cohort III receiving 3 doses of RotaTeq™/placebo. The primary investigator and the Ethics Review Committee will review blinded safety data and make decision based on their best clinical judgment to move study forward between cohorts. Duration for the entire study will be approximately 6-9 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ages 19 to 47 years for Cohort I
* Healthy children ages 2 to 6 years for Cohort II
* Healthy infants ages 6 to 12 weeks for Cohort III
* Negative pregnancy test for females in Cohort I
* Signed Informed Consent Forms (ICFs)

Exclusion Criteria:

* Participants in Cohorts I and II receiving any vaccine 14 days before or anticipated after study vaccine
* Participants in Cohort III receiving non-concomitant live vaccines 14 days before or after study vaccine
* Prior administration of any rotavirus vaccine
* Elevated temperature, with axillary temperature ≥37.1 Degrees C 24 hours before study vaccine
* Prior or active gastrointestinal illnesses, immunodeficiency
* Any condition which may interfere with evaluation of study objectives or make participation in the study unsafe for the participant

Ages: 6 Weeks to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 144 participants were enrolled; 48 in each of 3 cohorts. This study was conducted sequentially in the 3 different Cohorts, Chinese adults (Cohort I) first, followed by children (Cohort II), and then infants (Cohort III).
Period: Overall Study
Arm/Group | Cohort I - RotaTeq™, Adults | Cohort I - Placebo, Adults | Cohort II - RotaTeq™, Children | Cohort II - Placebo, Children | Cohort III - RotaTeq™, Infants | Cohort III - Placebo, Infants
Started | 24 | 24 | 24 | 24 | 24 | 24
Completed | 24 | 24 | 24 | 24 | 22 (One participant received placebo at the second dose in error, but completed the study.) | 20
Not Completed | 0 | 0 | 0 | 0 | 2 | 4
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 2 | 3
Not completed — Serious Adverse Event | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I - RotaTeq™, Adults | Cohort I - Placebo, Adults | Cohort II - RotaTeq™, Children | Cohort II - Placebo, Children | Cohort III - RotaTeq™, Infants | Cohort III - Placebo, Infants | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 144
Age, Customized [Number; unit: participants] — The inclusion criterion for Cohort I (adults) in this study was 19-47 years. However, one participant who was 49 years at study entry was randomized.
  participants
    6 weeks to 12 weeks (infants) | 0 | 0 | 0 | 0 | 24 | 24 | 48
    2 years to 5 years (children) | 0 | 0 | 24 | 24 | 0 | 0 | 48
    19 years to 49 years (adults) | 24 | 24 | 0 | 0 | 0 | 0 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 10 | 11 | 8 | 11 | 70
  Male | 11 | 7 | 14 | 13 | 16 | 13 | 74
Region of Enrollment [Number; unit: participants]
  China | 24 | 24 | 24 | 24 | 24 | 24 | 144

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: All serious adverse events (SAEs) were collected for 14 days following each dose to obtain the number of participants with serious adverse events.
Time Frame: up to 14 days post vaccination
Measure: Number; unit: Participants
Arm/Group | Cohort I - RotaTeq™, Adults | Cohort I - Placebo, Adults | Cohort II - RotaTeq™, Children | Cohort II - Placebo, Children | Cohort III - RotaTeq™, Infants | Cohort III - Placebo, Infants
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 3

2. Primary Outcome: Number of Serious Adverse Events
Description: The total number of serious adverse experiences (events) in participants up to 14 days post vaccination.
Time Frame: 14 days post vaccination
Measure: Number; unit: Events
Arm/Group | Cohort I - RotaTeq™, Adults | Cohort I - Placebo, Adults | Cohort II - RotaTeq™, Children | Cohort II - Placebo, Children | Cohort III - RotaTeq™, Infants | Cohort III - Placebo, Infants
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24
Events | 0 | 0 | 0 | 0 | 0 | 4

3. Secondary Outcome: Number of Infants With Fecal Vaccine Virus Shedding
Description: Fecal shedding of vaccine rotavirus in Cohort III (infants) was evaluated by determining the number of participants whose stool was positive by both (1) the Enzyme-linked Immunosorbent Assay (EIA) to detect the rotavirus antigen, and (2) PCR VP6 Genotyping (a polymerase chain reaction assay specific for rotavirus genome 6, coding for the VP6 protein of the vaccine virus). For analysis, two stool samples were collected per participant on separate days between Day 3 and Day 7 following each vaccination dose.
Time Frame: Between Day 3 and Day 7 following each of 3 doses of RotaTeq™/placebo
Population: Only participants in Cohort III, infants that received the scheduled dose of vaccination, and for whom the stool samples were available for testing, were included in the analysis for that dose.
Measure: Number; unit: Participants
Arm/Group | Cohort III - RotaTeq™, Infants | Cohort III - Placebo, Infants
Number analyzed (Participants) | 24 | 24
Participants
  Postdose 1 (n=23 for RotaTeq™, n=24 for placebo) | 3 | 0
  Postdose 2 (n=21 for RotaTeq™, n=22 for placebo) | 2 | 0
  Postdose 3 (n=22 for RotaTeq™, n=20 for placebo) | 3 | 0

ADVERSE EVENTS:
Description: One participant in the Cohort III-RotaTeq™ treatment group received RotaTeq™ at the first and third dose but placebo at the second dose in error. The participant had moderate or mild diarrhea after the second and third doses, respectively. The participant's AE data is included in the AE tables under the Cohort III-RotaTeq™ treatment group.
Arm/Group | Cohort I - RotaTeq™, Adults | Cohort I - Placebo, Adults | Cohort II - RotaTeq™, Children | Cohort II - Placebo, Children | Cohort III - RotaTeq™, Infants | Cohort III - Placebo, Infants
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 3/24
Other Adverse Events (participants affected / at risk) | 6/24 | 2/24 | 6/24 | 3/24 | 18/24 | 14/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I - RotaTeq™, Adults (N=24) | Cohort I - Placebo, Adults (N=24) | Cohort II - RotaTeq™, Children (N=24) | Cohort II - Placebo, Children (N=24) | Cohort III - RotaTeq™, Infants (N=24) | Cohort III - Placebo, Infants (N=24)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ENCEPHALITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I - RotaTeq™, Adults (N=24) | Cohort I - Placebo, Adults (N=24) | Cohort II - RotaTeq™, Children (N=24) | Cohort II - Placebo, Children (N=24) | Cohort III - RotaTeq™, Infants (N=24) | Cohort III - Placebo, Infants (N=24)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 13 (23) | 8 (19)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 9 (22) | 12 (25)
MALAISE (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 9 (11) | 5 (8)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (4)
HEADACHE (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/ presentation. SPONSOR review can be expedited to meet publication guidelines.